CLINICAL TRIAL: NCT06972472
Title: A Master Protocol to Investigate the Efficacy and Safety of Orforglipron Tablet Once Daily Compared With Placebo in Participants With Obesity or Overweight With and Without Type 2 Diabetes
Brief Title: A Study of Orforglipron (LY3502970) in Participants With Obesity or Overweight and Type 2 Diabetes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27362; 2025-521098-14-00 (EU CTIS Number); J2A-MC-GZP2 (Other: Eli Lilly and Company); J2A-MC-GZPO (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Overweight; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2 | interventions — orforglipron

STUDY DESIGN:
Intervention Model Description: Phase 3b
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Orforglipron Dose 1 (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Orforglipron Dose 2 (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Orforglipron Dose 3 (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Orforglipron Dose 4 (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970
  Arms: Orforglipron Dose 1; Orforglipron Dose 2; Orforglipron Dose 3; Orforglipron Dose 4
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to see how orforglipron, compared with placebo, helps improve glycemic control in participants with obesity or with overweight and type 2 diabetes. This trial is part of the master protocol study J2A-MC-GZPO.

Participation in the study will last about 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Have body mass index (BMI) ≥25 kilograms per square meter (kg/m2) at screening
* Have type 2 diabetes
* Have hemoglobin A1c (HbA1c) ≥7% and ≤10% at screening
* Have a history of at least one unsuccessful dietary effort to lose body weight

Exclusion Criteria:

* Have type 1 diabetes
* Have an unstable body weight within 90 days prior to screening
* Have New York Heart Association functional classification IV congestive heart failure or an acute cardiovascular condition within 90 days prior to screening
* Have acute or chronic hepatitis or pancreatitis
* Are taking other medications or alternative remedies to manage weight loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 40

SECONDARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline up to 72 weeks
Change from Baseline in HbA1c at Week 72 | Baseline, Week 72
Change from Baseline in Fasting Glucose | Baseline up to 72 weeks
Percentage of Participants Achieving HbA1c of <7.0% | Baseline up to 72 weeks
Percentage of Participants Achieving Weight Reduction of ≥5% | Baseline up to 72 weeks
Change from Baseline in Waist Circumference | Baseline up to 72 weeks
Change from Baseline in Body Max Index (BMI) | Baseline, Week 72
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline up to 72 weeks
Percent Change from Baseline in Triglycerides | Baseline up to 72 weeks
Change from Baseline in EQ-5D-5L | Baseline, Week 72
Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve (AUC-ss) of Orforglipron | Predose through Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (77):
- United States (32):
  - Clinical Research Institute of Arizona (CRI) - Sun City West, Sun City West, Arizona
  - Novak Clinical Research - Tucson - North La Cholla Boulevard, Tucson, Arizona
  - Norcal Endocrinology & Internal Medicine, San Ramon, California
  - Southern California Clinical Research, Santa Ana, California
  - Care Access - Thousand Oaks, Thousand Oaks, California
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - Innovation Medical Research Center - Fort Lauderdale, Fort Lauderdale, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Encore Medical Research, Hollywood, Florida
  - West Orange Endocrinology P.A., Ocoee, Florida
  - Care Access - Tampa, Tampa, Florida
  - Accel Research Sites - NeuroStudies Clinical Research Unit, Decatur, Georgia
  - Care Access - Decatur, Decatur, Georgia
  - Javara - Privia Medical Group Georgia - Savannah, Savannah, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Care Access - New Iberia, New Iberia, Louisiana
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Javara - Privia Medical Group - Silver Spring, Silver Spring, Maryland
  - Boeson Research MSO, Missoula, Montana
  - Javara - Nevada Health Centers - Carson City, Carson City, Nevada
  - The Machuca Foundation, Las Vegas, Nevada
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Javara - Tryon Medical Partners, Charlotte, North Carolina
  - Care Access - Fayetteville, Fayetteville, North Carolina
  - The Corvallis Clinic, P.C., Corvallis, Oregon
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Texas Valley Clinical Research (TVCR) - Mission, Mission, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
- Argentina (6):
  - CARE - Centro de Alergia y Enfermedades Respiratorias, Buenos Aires
  - CIPREC, Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Instituto Centenario, CABA
  - Instituto Médico Catamarca IMEC, Rosario
  - Centro de Diagnóstico y Rehabilitación (CEDIR), Santa Fe
- China (12):
  - Xuanwu Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - The Second Affiliated Hospital Chongqing Medical University, Chongqing
  - Zhujiang Hospital, Guangzhou
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - The Second People's Hospital of Hefei, Hefei
  - Jinan Central Hospital, Jinan
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Zhongda Hospital Southeast University, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - The Second Hospital of Tianjin Medical University, Tianjin
- Czechia (5):
  - MUDr. Alena Vachova, České Budějovice
  - Nemocnice Cesky Krumlov, Český Krumlov
  - VASOMED Clinic, Ostrava
  - Milan Kvapil s.r.o., Diabetologicka ambulance, Prague
  - Medical Plus, Uherské Hradiště
- Germany (7):
  - InnoDiab Forschung Gmbh, Essen
  - Medizentrum Essen Borbeck, Essen
  - Diabetes Zentrum Wilhelmsburg, Hamburg
  - AmBeNet GmbH, Leipzig
  - Gemeinschaftspraxis Dr. Taeschner/Dr. Bonigut, Leipzig
  - Medicover Neuroendokrinologie, Munich
  - RED-Institut GmbH, Oldenburg
- Japan (13):
  - Hasegawa Medicine Clinic, Chitose
  - The Institute of Medical Science, Asahi Life Foundation, Chūōku
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Fukuwa Clinic, Chūōku
  - Tokuyama Clinic, Mihama-ku,Chiba City
  - Medical Corporation Heishinkai ToCROM Clinic, Shinjuku-ku
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi
  - Olive Takamatsu Medical Clinic, Takamatsu
  - Shimokitazawa Tomo Clinic, Tokyo
  - Tsuchiura Medical & Health Care Center, Tsuchiura
  - Noritake Clinic, Ushiku
  - Medical Corporation Yuga Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi
  - Yokohama Minoru Clinic, Yokohama
- Puerto Rico (2):
  - Puerto Rico Health and Wellness Institute, Dorado
  - Isis Clinical Research Center, Guaynabo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Orforglipron (LY3502970) in Participants With Obesity or Overweight and Type 2 Diabetes (GZPO) — https://trials.lilly.com/en-US/trial/609395